CLINICAL TRIAL: NCT05038748
Title: A Pilot Study of Microbiome in Patients With Autism Spectrum Disorder and Their Unaffected
Brief Title: A Pilot Study of Microbiome in Patients With Autism Spectrum Disorder and Their Unaffected Siblings
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201810048RIND
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5 g of stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASD group: 80 youths with the clinical diagnosis of ASD according to the DSM-5 diagnostic criteria
  Interventions: Other: Psychiatric diagnosis; Other: ASD diagnosis
- Sibling group: 30 unaffected siblings of ASD youths
  Interventions: Other: Psychiatric diagnosis
- TD group: 40 healthy typical developing(TD) control from cohort established at Department of Psychiatry, National Taiwan University Hospital (NTUH) starting from 2007
  Interventions: Other: Psychiatric diagnosis

INTERVENTIONS:
Other: Psychiatric diagnosis — Kiddie Schedule for Affective Disorders & Schizophrenia (K-SADS) for DSM-5
Other: ASD diagnosis — Autism Diagnostic Interview-revised (ADI-R) and Autism Diagnostic Observation Scale (ADOS)
  Groups: ASD group

SUMMARY:
The primary aims are to identify important gut microbiota signatures for youth with ASD, to identify dysbiosis features for different levels of ASD features and clinical courses, to search the possibility to intervene the disease course if we can tease out the dysbiosis responsible for the flare-up and improvement of the symptoms of the disease. The secondary aims are to identify the clinical and neuropsychological measures that are associated with direct and indirect regulation or interactions from gut-brain axis signaling, and based our preliminary results on reducing the measures for future large-scale microbiome study in ASD.

DETAILED DESCRIPTION:
Background: Despite increased public awareness of autism spectrum d isorder (ASD) and extensive research on this neurodevelopmental disorder in the past decades, the underlying mechanisms of ASD remain unclear, and ASD is still recognized as having the highest disease and care burden among child psychiatric disorders regarding its long-term impairment across the lifespan. Hence, identifying the biomarkers for early detection and effective biological treatments for ASD is among the most challenging tasks all over the world. The concerns about physical comorbidities such as immune dysregulation, allergy, and gastrointestinal issues, etc. emerged in the recent decade. Hence, the new perspective of searching for the underlying mechanism for ASD also targets the associations between microbiota and ASD. However, despite many microbiome studies in ASD, they provided limited knowledge about the specific link that particular imbalance gut bacteria could affect the behavioral deficits in ASD because lack of consideration of the clinical and genetic heterogeneity of ASD. With only a few studies examining the well-defined ASD-related impairments, the GI system dysfunction, and the microbiomes, the associations among ASD-related symptoms, GI symptoms, and microbiota remain indistinct. Therefore, the investigators propose this pilot study to fill the gap between the potential role of microbiome as a biomarker for ASD to facilitate developing the treatment for ASD.

Method and material: The case-sibling control study design will be used to investigate microbiome in 60 probands with ASD, aged 7-25 yrs old, and 30 unaffected siblings either from the PI Gau's ASD cohort or the Department of Psychiatry, National Taiwan University Hospital. The parents of all the subjects will receive the Autism Diagnostic Interview-Revised (ADI-R) interviews and report on the questionnaires regarding autistic symptoms, emotional/behavioral problems, social functions, G-I symptoms, and life quality. The ASD and sibling subjects will receive the Autism Diagnostic Observation Scale and neuropsychological tasks. The experiment of microbiome will be conducted by the core lab of microbiome (co-PI Ni) at the college of medicine, National Taiwan University. The data analyses will combine microbiomics and the extensive behaviors/cognitive function variables to establish an objective potential pipeline.

Anticipated outcome: With the accomplishment of this project, the investigators will establish the comprehensive yet fewer bios for the ASD risk bio-factors in Asia, and provide the potential clinical interview and assessments related to GI symptoms regulated by microbiota. The potential biomarkers may be further used to developing the treatment for ASD.

Significance: Several features of this project constitute its significance: a wealth of measures of ASD phenotypes (valid phenotype), ASD as a catastrophic disease (importance), the first ASD study with unaffected sibling design for microbiomics studies in ASD (originality), and new approaches and technologies (novelty) for searching microbiomics in ASD.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of ASD defined by the DSM-IV confirmed by ADI-R or ADOS and also clinical reappraisal based on the newly release DSM-5 criteria for ASD
* ages range from 7 to 25 at the time now
* at least one biological parent
* parents that are both Han Chinese in Taiwan

Exclusion Criteria:

* intellectual disability
* epilepsy
* ADHD
* autoimmune diseases

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The cohort was established at the Department of Psychiatry, National Taiwan University Hospital (NTUH) starting from 2007.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Autism Diagnostic Interview-Revised (ADI-R) | 1 hour
  Including reciprocal social interaction, communication, and repetitive behaviors and stereotyped patterns, for children with a mental age from about 18 months into adulthood. The coding of some items is converted to numeric scores "0" if no evidence of abnormality exists, "1" if some evidence of abnormality exists, and "2" if evidence of marked abnormality. Higher scores mean more severe clinical deficits.
Autism Diagnostic Observation Scale (ADOS) | 1 hour
  Including communication, social interaction, creativity, stereotyped behaviors and restricted interests. The coding of some items is converted to numeric scores "0" if no evidence of abnormality exists, "1" if some evidence of abnormality exists, and "2" if evidence of marked abnormality. Higher scores mean more severe clinical deficits.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan